CLINICAL TRIAL: NCT00003746
Title: Daily Versus Weekly Administration of 2-Chlorodeoxyadenosine (CDA) in Patients With Hairy Cell Leukemia
Brief Title: Daily or Weekly Cladribine in Treating Patients With Hairy Cell Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 32/98; SWS-SAKK-32/98; EU-98074
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Prolymphocytic | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDA day (Active Comparator): CDA:0.14 mg/kg/day Bolus s.c. (standard) days 1-5
  Interventions: Drug: 2-chlorodeoxyadenosine (CDA) daily
- CDA week (Active Comparator): CDA:0.14 mg/kg/week Bolus s.c. weeks 1-5
  Interventions: Drug: 2-chlorodeoxyadenosine weekly

INTERVENTIONS:
Drug: 2-chlorodeoxyadenosine (CDA) daily — Daily administration
  Arms: CDA day
Drug: 2-chlorodeoxyadenosine weekly — Weekly administration
  Arms: CDA week

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if giving cladribine once a day is more effective than giving cladribine once a week in patients with hairy cell leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of cladribine given once a day to cladribine given once a week in treating patients with hairy cell leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the acute hematotoxicity and infection rate with daily and weekly administration of cladribine in patients with hairy cell leukemia.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive daily subcutaneous bolus injections of cladribine (2-CDA) for 5 days (standard dose).
* Arm II: Patients receive weekly subcutaneous bolus injections of 2-CDA for 5 weeks.

Patients showing complete or partial remission at evaluation on day 71 of the first treatment course do not receive any further treatment until relapse or disease progression is evident.

Patients showing minor or no response on day 71 of the first treatment course receive a subsequent course of standard dose 2-CDA.

Patients are followed every 3 months for 2 years, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classic form or prolymphocytic variant hairy cell leukemia (HCL)
* Newly diagnosed HCL or progressive disease after prior treatment

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* NCI 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.3 mg/dL

Other:

* HIV negative
* Not pregnant
* No other prior or concurrent malignancy except carcinoma in situ of the cervix or basal or squamous cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since any prior therapy and recovered

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent cytoreductive therapy
* No prior cladribine

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1998-09; Primary Completion 2005-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Acute hematotoxicity at 10 weeks following study treatment | 10 weeks
Acute infection rate at 10 weeks following study treatment | 10 weeks

SECONDARY OUTCOMES:
Hospital admission frequency and length at 10 weeks following study treatment | 10 weeks
Blood support at 10 weeks following study treatment | 10 weeks
Remission rate | 10 weeks
Remission duration | 10 weeks
Relapse-free survival | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Zenhaeusern, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- [Result] Zenhausern R, Schmitz SF, Solenthaler M, Heim D, Meyer-Monard S, Hess U, Leoncini L, Bargetzi M, Rufener B, Tobler A. Randomized trial of daily versus weekly administration of 2-chlorodeoxyadenosine in patients with hairy cell leukemia: a multicenter phase III trial (SAKK 32/98). Leuk Lymphoma. 2009 Sep;50(9):1501-11. doi: 10.1080/10428190903131755. PMID 19672771